CLINICAL TRIAL: NCT02733874
Title: A Trial That Compound Clobetasol Propionate Ointment Treats Patients With Mild to Moderate Psoriasis Vulgaris.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Professor, doctoral tutor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZY2015001
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- test group (Experimental): Compound Clobetasol Propionate Ointment
  Interventions: Drug: Compound Clobetasol Propionate Ointment
- control group (Active Comparator): Calcipotriol Betamethasone Ointment
  Interventions: Drug: Calcipotriol Betamethasone Ointment

INTERVENTIONS:
Drug: Compound Clobetasol Propionate Ointment
  Arms: test group
Drug: Calcipotriol Betamethasone Ointment
  Arms: control group

SUMMARY:
A multi-center, randomized, single blind, positive controlled trials that assess the effectiveness, safety and cost-effectiveness analysis in patients with mild to moderate psoriasis vulgaris and compare Compound Clobetasol Propionate Ointment to Calcipotriol Betamethasone Ointment.

Objectives of Study：

1. Compare Compound Clobetasol Propionate Ointment to Calcipotriol Betamethasone Ointment in the treatment of mild to moderate psoriasis vulgaris in effectiveness and safety;
2. Compare the cost-effectiveness analysis of two treatment programs.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent has been signed in;
2. Patients who were 18~65 years of age, stable psoriasis patients, the gender is not limited;
3. The lesion area does not exceed 10% of the total surface area of the body;
4. The overall evaluation of the researchers (Physician Global Assessment,PGA) greater than or equal to 2;
5. The observation of target lesions of minimum diameter greater than or equal to 2cm.

Exclusion Criteria:

1. Patients who have known or been doubted of being allergic to the composition of the drug;
2. Patients who were diagnosed as non-psoriasis vulgaris (such as erythrodermic type, pustular psoriasis, arthritis), and developing psoriasis vulgaris;
3. Patients who have illnesses in severe central nervous system, cardiovascular system, kidney, liver, digestive tract, respiratory system, metabolism and skeletal muscle system and mental disorders;
4. Patients with other diseases may affect the assessment of efficacy, such as eczema, etc.;
5. Liver functions(such as Alanine aminotransferase, Aspartate transaminase) is 2 times greater than(or equal to) the upper limit of normal value, or renal functions (such as creatinine) is 1.5 times greater than(or equal to) the upper limit of normal value;
6. Patients with hypercalcemia whose serum calcium values exceed the upper limit of the normal value or patients who were suspected of having a disease of hypercalcemia;
7. Patients who are taking drugs that affect metabolism of calcium. Drugs that increase the serum calcium values: agents containing calcium, active vitamin D3 medication, injection, anabolic agents (ipriflavone preparations); Drugs that decrease the serum calcium values: calcitonin preparation, double phosphate ester compound preparation, sex hormone preparations).
8. Patients who were randomly divided into groups had received systemic biological treatment (listed or unlisted), such as: ustekinumab treatment accepted by patients after the past 12 weeks, infliximab, adalimumab treatment accepted by patients after the past 8 weeks, infliximab, etanercept treatment accepted by patients after the past 4 weeks accepted and so on;
9. Patients who have accepted non-abiotic systemic therapy that may have an effect on psoriasis, including but not limited to vitamin A preparations, cortical hormone, vitamin D analogs, immunosuppressant, compound glycyrrhizin, traditional Chinese medicine and so on after the past 4 weeks of random entry or test period.
10. Patients who have were accepted psoralen ultraviolet A(PUVA) treatment after the past 4 weeks of random entry or test period.
11. Patients who have accepted ultraviolet therapy or partial treatments of psoriasis drugs after the past 2 weeks of random entry or test period;
12. Patients who have used concomitant drugs recently in the past 2 weeks after random entry or plan to use concomitant drugs during test period, such as Beta blockers, anti malaria drugs, lithium preparations, etc.;
13. Patients who have accepted other clinical trials after the the last 4 weeks of random entry;
14. Patients who work outside for a long time with sun exposure may have an impact on the diagnosis and treatment of the disease.
15. Women of lactation, pregnancy and childbearing age who refuse to accept effective contraceptive measures.
16. Patients who have known or been suspected of non-compliance, such as alcoholism, drug dependence or mental illness, etc, and can not be suitable to the clinical trials judged by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The improvement of psoriasis area and severity index scores(PASI scores) | At baseline, 2 weeks and 4 weeks after baseline.
  The improvement of psoriasis area and severity index scores(PASI scores) are a system that assesses the damage of psoriasis severity and treatment response . The system is used to classify and evaluate according to the severity of lesions, areas of skin lesion and body surface area ratio of various body parts.
The overall evaluation of the researchers (Physician Global Assessment,PGA) | At baseline, 2 weeks and 4 weeks after baseline.
  On every visiting viewpoint , researchers give a mark of the infiltration / hypertrophy (I), erythema (E) and scales (s) according to the level.PGA scores are acquired by the average of above three kinds of scores.
The Symptom score reduce index (SSRI) | 4 weeks after baseline.
  1)According to the improvement of psoriasis area and severity index scores(PASI scores) before and after treatments, the symptom score reduce index (SSRI) was calculated.
  2）The symptom score reduce index (SSRI) = (the PASI scores before treatment - the PASI scores after treatment) / the PASI scores before treatment x 100%
Efficiency of treatment | 4 weeks after baseline.
  1）Healing patients : SSRI ≥ 90%, Marked effectiveness patients : 60% < SSRI < 90%, Improvement patients : 20% < SSRI < 60%, ineffectiveness patients :SSRI < 20%.
  2)Efficiency of treatment = (The number of healing patients + The number of markedly effective patients + The number of improved patients ) / total number of patients in this group x 100%

SECONDARY OUTCOMES:
Healing rate | 4 weeks after treatment
  1）Healing patients : SSRI ≥ 90%, Marked effectiveness patients : 60% < SSRI < 90%, Improvement patients : 20% < SSRI < 60%, ineffectiveness patients :SSRI < 20%.
  2)Healing rate = The number of healing patients / total number of patients in this group x 100%
Markedly effective rate | 4 weeks after treatment
  1）Healing patients : SSRI ≥ 90%, Marked effectiveness patients : 60% < SSRI < 90%, Improvement patients : 20% < SSRI < 60%, ineffectiveness patients :SSRI < 20%.
  2)Markedly effective rate = The number of markedly effective patients / total number of patients in this group x 100%
Response rate of PASI (PASI 75) after the treatment of 4 weeks | 4 weeks after treatment
  Response rate of PASI (PASI 75) after the treatment of 4 weeks = The number of patients whose SSRI are more than 75% / total number of patients x 100%
Response rate of PGA ( basic fading rate of PGA) after the treatment of 4 weeks | 4 weeks after treatment
  Response rate of PGA ( basic fading rate of PGA) after the treatment of 4 weeks：patients with 1 score of PGA for the last time/ total number of patients in this group x 100%